CLINICAL TRIAL: NCT05212636
Title: Using Repetitive Transcranial Magnetic Stimulation to Study the Role of Frontostriatal Circuit in Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Po-See, Chen, Principal Investigator, Professor, Visiting Staff Psychiatrist of Department of Psychiatry, Professor (joint appointment) of Institute of Behavioral Medicine, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-108-092
Record Dates: First submitted 2021-10-07; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Depressive Disorder, Major
Keywords: Repetitive Transcranial Magnetic Stimulation (rTMS); Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDD patient with HRSD score of at least 18 (Experimental): MDD patients who meet the DSM-5 diagnostic criteria of MDD and their current episode show a 17-Item Hamilton Rating Scale for Depression (HRSD) score of at least 18
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — A total of 12 sessions of rTMS (5 sessions per week for 2 weeks, follow by 1 session per week for next 2 weeks) .
  Other Names: Antidepressants

SUMMARY:
Major depressive disorder (MDD) is a common, severe, and often life-threatening illness that involves the body, mood, and thoughts. The natural course of MDD tends to worsen without treatment, while people with MDD can lead healthy and productive lives when the illness is effectively treated. Up to 50% of the patients show no response to current available antidepressants.Two major non-invasive brain stimulation (NIBS) tools have been applied for the treatment of psychiatric diseases so far, transcranial magnetic and direct current stimulation (TMS, tDCS). TMS induces a strong magnetic field (magnetic pulses) through the skull into the brain, which generates electrical currents in brain tissue and induces neuronal firing, leading to after-effects, i.e. neuroplasticity, eventually. Neuronal effects of rTMS has been proven to last beyond the actual time of stimulation, enabling altered brain activity for an extended period of time. Adding on rTMS treatment could even give a chance to treat the physical comorbidities and enhance cognitive function in MDD. Nevertheless, underlying neurobiological mechanism of rTMS treatment remains unclear. Reports showed chronic psychosocial stressors are associated with altered frontal-striatal circuitry activation and connectivity. Indeed, aberrant fronto-striatal connectivity and reduced sustain fronto-striatal activation were noticed in MDD patients. However, the specific correlations between fronto-striatal connectivity changes and rTMS treatment outcomes in MDD remain unclear. In this study fMRI will be used to measure the possible correlations between the fronto-striatal circuit activation / connectivity with (1) mood symptoms presentations, (2) neurocognitive measurements, (3) HPA and ANS activities, and (4) immune and metabolic status (cytokines, adipokines and insulin levels) in patients with MDD. Then the possible changes in fronto-striatal FC over a four-week treatment course with 10 Hz rTMS stimulation to left dorsolateral prefrontal cortex will be measured. The FC changes will be tested to find out whether correlate with treatment outcomes, HPA and ANS activity; and immune/metabolic indices changes.

We hypothesize that rTMS as an add-on therapy would change the fronto-striatal FC that correlated with mood symptom improvement, neurocognitive measurements, HPA and ANS activity, inflammatory and metabolic homeostasis in patients with MDD.

DETAILED DESCRIPTION:
BACKGROUNDＡND SIGNIFICANCE:

1. The scale of the global impact of MDD is substantial, with mental illness constituting an estimated 7.4% of the world's measurable burden of disease. With a period of sustained disruption of mood, patients with MDD have the symptoms of distortions in perception and somatic functioning, and impairment in social functioning. Among the possible comorbidities, epidemiologic evidences have indicated increased risk of metabolic disturbances in MDD patients. The metabolic disturbances are correlated with higher morbidity and mortality in patients with MDD. Comorbid diabetes and MDD are a major clinical challenge as the outcomes of both conditions are worsened by the other.
2. Although there are several types of antidepressant medications used to treat depressive disorders, up to 50% of the patients do not show response to antidepressants treatment. Importantly, increased inflammasome activation, cognitive impairment, and insulin resistance follow the non-remitting and recurrence in treating MDD, and might further dampen antidepressant treatment response. Moreover, the systemic effect of antidepressants treatment has linked to increased risk of metabolic disturbance.

   Recently, the development of non-invasive brain stimulation (NIBS) has provided alternative therapeutic options for psychiatric disorders. Two major NIBS tools have been applied for the treatment of psychiatric diseases so far, transcranial magnetic and direct current stimulation (TMS, tDCS). TMS includes induction of a strong magnetic field (magnetic pulses) through the skull into the brain. The magnetic pulses generate electrical currents in brain tissue and consequently induce neuronal firing. Repetitive TMS (rTMS) induces after-effects of the intervention, i.e. neuroplasticity. In general, low frequency (<1 Hz) rTMS reduces neuronal activity and cortical excitability, while higher frequency (>5 Hz) rTMS results in excitability enhancement. Neuronal effects of rTMS been proven to last beyond the actual time of stimulation, enabling altered brain activity for an extended period of time. The rTMS has emerged as a promising alternative strategy for treatment-resistant depression; however, the underlying neurobiological mechanisms are still not fully understood. In addition, adding on rTMS treatment could give a chance to treating the physical comorbidities and enhance cognitive function in MDD. The incorporation of biological assessments into future rTMS clinical studies will help in this regard.
3. The frontal-striatal circuits mediate broadly dissociable cognitive and behavioural processes through limbic (ventromedial prefrontal regions, ventral striatum - VS, ventral tegmental area - VTA), motor (supplementary motor areas - SMAs, putamen, substantia nigra) and cognitive (lateral prefrontal and caudate) functional connectivity (FC). Reports had showed chronic psychosocial stressors are associated with altered frontal-striatal circuitry activation and connectivity. Structure and functional abnormalities of the striatum and frontal cortex have been reported consistently in studies in mood disorders. In MDD, patients are characterized by aberrant fronto-striatal connectivity and reduced sustain fronto-striatal activation. The MDD related executive dysfunction also showed clinical presentations and neuroimaging findings consistent with frontal-striatal circuitry abnormalities. Within the circuit, striatum is associated with reward and motor processing systems and receives emotion-related information and motivation from the frontal lobe, anterior cingulate cortex, and amygdala. The high incidence of depressive symptomatology following left frontal and basal ganglia lesions also implicate their roles in MDD.

   The dysfunctional fronto-striatal circuits also link to the metabolic comorbidities and cognitive deficits, that involved executive functioning, attention, processing speed, and working memory in patients with mood disorders. Regarding metabolic control, the fronto-striatal functional connectivity changes affect food craving. And the altered reciprocal loop from the medial prefrontal cortex could promote overeating and metabolic disturbance. Moreover, animal and clinical studies had suggested that striatal dopamine signaling plays a role in systemic glucose regulation. On the opposite, brain circuitry connectivity could be enhanced by either glucose loading or insulin challenge. Moreover, insulin resistance related aberrant functional circuitry has been demonstrated in patients with type 2 diabetes. Individuals with insulin resistance also showed aberrant fronto-striatal connectivity with failure to shift from reward toward cognitive control circuit.
4. Changes in the ability to sustain fronto-striatal connectivity during the regulation of positive affect are associated with gains in positive affect through anti-depressants treatment. Duloxetine has been noted to modulate the FC between striatum and dorsolateral prefrontal cortex while showing symptomatic improvement. Moreover, the fronto-striatal connectivity attenuation among reward-processing regions could predict response to psychotherapy in MDD. Therefore, the degree of connectivity within the fronto-striatal circuit has been considered as a predictive biomarker of remission in treating MDD. Changes in FC might also relate to outcome of rTMS treatment of MDD. The FC variations represent the mechanism of action of rTMS and explain the individual difference in treatment outcome. However, the specific correlations between fronto-striatal connectivity changes and rTMS treatment outcomes in MDD remain unclear.

By using fMRI, in this project we will first measure the possible correlations between the fronto-striatal circuit activation/connectivity with (1) mood symptoms presentations, (2) neurocognitive measurements, (3) HPA and ANS activities, and (4) immune and metabolic status (cytokines, adipokines and insulin levels) in patients with MDD. Then we will measure the possible changes in fronto-striatal FC over a four-week treatment course with 10 Hz rTMS stimulation to left dorsolateral prefrontal cortex. We will test if the FC changes correlate with treatment outcomes, HPA and ANS activity; and immune/metabolic indices changes.

HYPOTHESIS:

We hypothesize that rTMS as an add-on therapy would change the fronto-striatal FC that correlated with mood symptom improvement, neurocognitive measurements, HPA and ANS activity, inflammatory and metabolic homeostasis in patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

* meet the DSM-5 diagnostic criteria and their current episode show a 17-item Hamilton Rating Scale for Depression (HRSD-17) score of at least 18
* show no clinical response to an adequate dose of an antidepressant
* could not tolerate at least two antidepressants in the current episode will be enrolled consecutively by trained psychiatrists
* Patients should receive a stable antidepressant regimen for at least 4 weeks before screening and continue during treatment

Exclusion Criteria:

* had DSM-5 diagnosis for substance abuse within the past three months
* had taken monoamine oxidase inhibitors
* had an organic mental disorder, mental retardation, dementia, or other diagnosed neurological illness
* had a surgical condition or a major physical illness
* underwent course of electroconvulsive therapy (ECT) within the last three months
* the presence of a cardiac pacemaker, intracranial implant, or metal in the cranium
* taking any anticonvulsant or if more than three adequate antidepressant trials had failed (determined by antidepressant treatment history form).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Mood Symptom Severity at Numerous Timepoints within 3 Months Period | Week 0, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12.
  Evaluation for disease severity by using the 17-item Hamilton Rating Scale for Depression (HAM-D) by trained senior psychiatrists. The same rater administers the scale for each patient. Higher scores represent worse mood symptoms.
Iowa gambling task (IGT) with Functional MR Imaging | Week 0
  The subject will be asked to turn a card from 4-decks voluntarily, and maximize gains and minimize losses during the game.
Change from Baseline homeostasis model assessment-estimated insulin resistance (HOMA-IR) index at Numerous Timepoints within 3 Months | Week 0, Week 4, Week 8, Week 12
  The homeostasis model assessment-estimated insulin resistance (HOMA-IR) index is calculated as the product of the fasting plasma insulin level (uIn/ml) and the fasting plasma glucose level (mg/dl), divided by 405. Insulin resistance is defined as HOMA-IR ≥2.5.
Change from Baseline Waist and Hip Circumference at Numerous Timepoints within 3 Months | Week 0, Week 4, Week 8, Week 12
  Waist and hip circumference (to the nearest 0.1 cm)
Change from Baseline Fasting Serum Leptin Level at Numerous Timepoints within 3 Months | Week 0, Week 4, Week 8, Week 12
  Measured using ELISA method (Linco Research, USA)
Change from Baseline Fasting Serum Lipid Level at Numerous Timepoints within 3 Months | Week 0, Week 4, Week 8, Week 12
  Fasting total cholesterol, high density lipoprotein cholesterol (HDL), low-density lipoprotein cholesterol (LDL) and triglyceride (TG) concentrations will be measured.
Change from Baseline Immunological Markers at Numerous Timepoints within 3 Months | Week 0, Week 2, Week 3, Week 4, Week 8, Week 12
  The fasting plasma CRP level will be assessed using an high-sensitivity CRP ELISA kit (Bender MedSystems, USA).
Change from Baseline Neurocognitive performance at 3 Months | Week 0, Week 12
  Neurocognitive performance will be assessed using Continuous Performance Test (CPT), Finger-Tapping Test (FTT) and Wisconsin Card-Sorting Test (WCST).

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan